CLINICAL TRIAL: NCT00004926
Title: A Phase I Study of Oral ILX23-7553 in Patients With Solid Tumors
Brief Title: ILX23-7553 in Treating Patients With Solid Tumors That Have Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-99078; CDR0000067610 (Registry Identifier: PDQ (Physician Data Query)); ILEX-VITD-101-A1; NCI-G00-1699
Record Dates: First submitted 2000-03-07; First posted 2004-03-16 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Ro 23-7553

INTERVENTIONS:
Dietary Supplement: vitamin D3 analogue ILX23-7553

SUMMARY:
RATIONALE: ILX23-7553 may help solid tumor cells develop into normal cells.

PURPOSE: Phase I trial to study the effectiveness of ILX23-7553 in treating patients who have solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and recommended phase II dose of ILX23-7553 in patients with refractory solid tumors. II. Determine the principal and dose limiting toxicities of this treatment regimen in terms of duration and reversibility in this patient population. III. Determine the preliminary evidence of antitumor activity with this treatment regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients receive oral ILX23-7553 for 5 days. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of ILX23-7553 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 or 2 of 10 patients experience dose limiting toxicity. Patients are followed monthly for at least 2 months.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor refractory to conventional therapy or for which no standard therapy exists Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL (regardless of liver metastases) SGOT/SGPT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Calcium no greater than 9.5 mg/dL No nephrocalcinosis Cardiovascular: No congestive heart failure No angina or ischemia Other: Ability to swallow or nasogastric or gastrostomy tube present Adequate organ and immune system function No known hypersensitivity to ILX23-7553 or analogues HIV negative No active uncontrolled infection No other severe disease or psychiatric disorder that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas or mitomycin) and recovered No concurrent curative antineoplastic drugs Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent curative radiotherapy Surgery: At least 4 weeks since prior surgery and recovered Other: At least 30 days since prior investigational agents At least 2 weeks since prior vitamin D, calcium supplementation, or cholestyramine No concurrent vitamin D, calcium supplementation, or cholestyramine No concurrent digoxin No concurrent hypercalcemia therapy (i.e., biphosphonates or insulin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2002-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Soignet, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - New Jersey Medical School, Newark, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York